CLINICAL TRIAL: NCT07109531
Title: A Randomized, Controlled, Open-Label, Multicenter, Phase 3 Study to Evaluate the Efficacy and Safety of ASKC202 in Combination With Limertinib Versus Platinum-based Chemotherapy in Participants With MET Amplification/Overexpression Locally Advanced or Metastatic NSCLC Who Have Failed After Prior EGFR-TKI Therapy.
Brief Title: ASKC202 Combined With Limertinib Versus Platinum-based Chemotherapy in Treatment of Locally Advanced or Metastatic NSCLC With MET Amplification/Overexpression After Failure of EGFR-TKI Therapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASKC202-301
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced or Metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, open-label, multicenter, phase 3 clinical study. The primary endpoint of this study is PFS as assessed by BIRC. patients with locally advanced or metastatic NSCLC with MET amplification/Overexpression after failure of EGFR inhibitor therapy are randomly assigned 1:1 stratified by MET amplification (MET GCN≥10 or MET GCN<10 )and brain metastasis (YES or NO) and EGFR mutation type(L858R；Del19) to receive ASKC202+ Limertinib or platinum-based chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASKC202 + Limertinib (Experimental): ASKC202+Limertinib
  Interventions: Drug: ASKC202+ Limertinib
- Pemetrexed + Cisplatin /Carboplatin (Active Comparator): Pemetrexed+Cisplatin/Carboplatin
  Interventions: Drug: Pemetrexed + Cisplatin /Carboplatin

INTERVENTIONS:
Drug: ASKC202+ Limertinib — ASKC202 orally once per day (QD) combined with Limertinib orally BID for every cycle of 21 days until disease progression or other criteria for treatment discontinuation will be met.
  Arms: ASKC202 + Limertinib
Drug: Pemetrexed + Cisplatin /Carboplatin — The standard chemotherapy treatment of cisplatin/carboplatin combined with pemetrexed on Day 1of 21 day cycles for 4~6 cycles (every 3 weeks).
  Arms: Pemetrexed + Cisplatin /Carboplatin

SUMMARY:
This study is designed to compare the safety and efficacy of ASKC202 combined with Limertinib Versus platinum-based chemotherapy in locally advanced or metastatic NSCLC With MET Amplification/Overexpression after disease progression on EGFR tyrosine kinase inhibitor.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, multicenter, phase 3 clinical study to valuate the efficacy and safety of ASKC202 combined with Limertinib in locally advanced or metastatic NSCLC with MET amplification/overexpression after failure of EGFR inhibitor therapy. Participants will continue to receive treatment until disease progression, intolerable toxicity, withdrawal of informed consent, death, or any other reasons for treatment discontinuation, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent;
2. Patients at least 18 years of age;
3. Locally advanced or metastatic non-small cell lung cancer (NSCLC);
4. Objective disease progression following prior EGFR-TKI therapy;
5. EGFR mutation with MET amplification/Overexpression by a central laboratory;
6. Measurable lesions based on RECIST 1. 1;
7. ECOG performance status 0 or 1;
8. Expected survival >12 weeks;
9. Adequate bone marrow reserve or organ function.

Exclusion Criteria:

1. Prior or ongoing treatment with any c-Met target;
2. Previously received systemic chemotherapy;
3. Patients requiring continuous use of systemic immunosuppressants or systemic corticosteroids within 2 weeks prior to the first dose.
4. Patients who underwent other major surgical procedures other than diagnosis or biopsy within 4 weeks prior to the first dose, or who were expected to undergo major surgeries during the study period;
5. Prior to the first administration, there are unhealed toxic reactions of ≥ grade 2 (CTCAE 5.0 standard) associated with any previous treatment, any level of hair loss, and platinum drugs Except for grade 2 neuropathy caused;
6. Patients with leptomeningeal metastasis, brainstem metastasis, or spinal cord compression;
7. Presence of dysphagia or gastrointestinal disorders that may interfere with oral medication absorption;
8. Previous history includes interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid therapy, or evidence of clinically active ILD；
9. Have previously received hematopoietic stem cell transplants or solid organ transplants, or plan to receive hematopoietic stem cell transplants or solid organ transplants during the current period of study;
10. There are serious or active infections that required intravenous antibiotics or hospitalization, such as HBV (HBsAg-positive and peripheral HBV-DNA titer test≥1×104 copies/mL or 2000 IU/mL), HCV, HIV, and syphilis;
11. Serious or uncontrolled cardiovascular disease;
12. Pregnant or lactating females;
13. Other primary malignancies have been diagnosed within the last 5 years, and the following conditions can be enrolled: non-melanoma skin cancer, superficial bladder cancer, cervical carcinoma in situ that has undergone surgery and has been cured;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) by BIRC | 2 years
  Progression-free survival (PFS) using BIRC assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).Progression-free survival was deﬁned as the time from date of randomization until the documentation of objective disease progression (PD) or death from any cause in the absence of progression (whichever occurred first).

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator | 2 years
  Progression-free survival (PFS) using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1).Progression-free survival was deﬁned as the time from date of randomization until the documentation of objective disease progression (PD) or death from any cause in the absence of progression (whichever occurred first).
Overall Survival (OS) | 3 years
  The time from the date of randomization to the date of death .
Objective Response Rate (ORR) | 2 years
  ORR was defined as the percentage of participants with complete response (CR) or partial response (PR) .
Disease Control Rate (DCR) | 2 years
  DCR was defined as the percentage of participants with complete response(CR), partial response(PR) and stable disease(SD).
Duration of Response (DoR) | 2 years
  Duration of response was defined as the time from when the criteria for CR or PR were first met to the occurrence of an objective disease progression or death.
Incidence and severity of treatment-emergent adverse events | 2 years
  Assessed by number and severity of adverse events as recorded on the case report form NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China